CLINICAL TRIAL: NCT03932201
Title: Observational Study Evaluating Effectiveness and Safety of Real-World Treatment With Damoctocog Alfa Pegol in Previously Treated Patients With Hemophilia A
Brief Title: Evaluating Effectiveness and Long Term Safety of Damoctocog Alfa Pegol in Patients, Who Have Been Diagnosed With Hemophilia A
Acronym: HEM-POWR
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20002
Record Dates: First submitted 2019-04-18; First posted 2019-04-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Previously treated patient (PTPs) with hemophilia A: Previously treated patients with hemophilia A receiving damoctocog alfa pegol with any kind of treatment modality (on-demand, prophylaxis, or intermittent prophylaxis)。
  Interventions: Drug: Damoctocog alfa pegol (Jivi, Bay94-9027)

INTERVENTIONS:
Drug: Damoctocog alfa pegol (Jivi, Bay94-9027) — Follow clinical practice. BAY94-9027 is a B-domain-deleted recombinant factor VIII (rFVIII) product site-specifically conjugated to a single (dual 30-kDa branched) 60-kDa polyethylene glycol (PEG) molecule. BAY 94-9027 is intended for prophylaxis and treatment of bleeds in patients with hemophilia A aged ≥12 years, with a narrow, predictable weekly dose that allows for the treatment regimen to be tailored to individual patient needs.

SUMMARY:
The aim of the HEM-POWR study is to understand better how Damoctocog alfa pegol (Jivi) is used to treat people with Hemophilia A in day-to-day life, how well the treatment is tolerated and how satisfied patients and physicians are with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A.
* Patients previously treated for Hemophilia A.
* Patients without previous history of inhibitors or patients with previous history of inhibitors on standard prophylaxis therapy for at least 1 year prior to study entry.
* No current evidence of FVIII inhibitor or clinical suspicion of FVIII inhibitor.
* Initiation of or currently on damoctocog alfa pegol with any kind of treatment modality (on-demand, prophylaxis, or intermittent prophylaxis).
* Signed informed consent/assent.

Exclusion Criteria:

* Concurrent participation in an investigational program with interventions outside of routine clinical practice.
* Diagnosis of any other bleeding/coagulation disorder other than hemophilia A.
* Contra-indications according to the local marketing authorization.
* Patient on immune tolerance induction (ITI) treatment at the time of enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously treated patients with hemophilia A receiving damoctocog alfa pegol with any kind of treatment modality (on-demand, prop hylaxis, or intermittent prophylaxis).
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean annualized number of reported total bleeds in patients with hemophilia A | Up to 36 months
Median annualized number of reported total bleeds in patients with hemophilia A | Up to 36 months

SECONDARY OUTCOMES:
Occurrence of AEs. | Up to 36 months
  Adverse Events (AEs) includes:
  AEs of special interest, Adverse Event, Serious Adverse Event, Adverse reaction.
  AEs of special interest includes: hypersensitivity reactions, loss of drug effect, renal impairment, neurocognitive disorders, inhibitor development.
Duration of AEs. | Up to 36 months
Treatment of AEs. | Up to 36 months
Severity of AEs. | Up to 36 months
Outcome of AEs. | Up to 36 months
Number of infusions and FVIII consumption to achieve hemostasis during surgery | Up to 36 months
Change in joint scores (HJHS) | From baseline to 12 months, 24 months and 36 months
  HJHS:Hemophilia Joint Health Score
Joint status evaluation by ultrasound (HEAD-US score), if available or part of standard clinical practice. | Up to 36 months
  HEAD-US:Hemophilia Early Arthropathy Detection with Ultrasound
Change of number of affected joints by patient | From baseline to 12 months, 24 months and 36 months
Annualized number of spontaneous, joint, and trauma bleeds | Up to 36 months
Number of reported bleeds during the study compared with number of reported bleeds for previous FVIII products in the 12 months prior to enrollment into the study. | Up to 36 months
  Bleeds includes total, spontaneous, joint, and trauma.
Proportion of patients with 0 bleeds, and the difference in proportion comparing to previous prophylaxis treatment. | Up to 36 months
AUC for previous FVIII products versus damoctocog alfa pegol. | Up to 36 months
  AUC:Area under the plasma concentration versus time curve
Half-life [t½] for previous FVIII products versus damoctocog alfa pegol. | Up to 36 months
FVIII trough for previous FVIII products versus damoctocog alfa pegol. | Up to 36 months
FVIII peak levels for previous FVIII products versus damoctocog alfa pegol. | Up to 36 months
In-vivo recovery for previous FVIII products versus damoctocog alfa pegol. | Up to 36 months
Number of infusions to control for a bleed | Up to 36 months
Changes of Hemo-SAT A score | From baseline to 12 months, 24 months and 36 months
  Hemo-SAT A:Hemophilia Treatment Satisfaction Questionnaire for adults。The Hemo-SAT questionnaire version for adults (Hemo-SAT A) consists of 34 items pertaining to 6 dimensions (Ease & Convenience, Efficacy, Burden, Specialist/Nurses, Center/Hospital, General Satisfaction).
Changes of Hemo-QoL (A and SF) score | From baseline to 12 months, 24 months and 36 months
  Hemo-QoL-A:Hemophilia Quality of Life Measure for adults Hemo-QoL-SF:Hemophilia Quality of Life short form for children Hemo-QoL-A is a hemophiliaspecific quality of life questionnaire for adults aged 18 years and above. The questionnaire has 41 items covering 6 domains: Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact, and Treatment Concerns. For patients younger than 18 years, the Hemo-QoL-SF Questionnaire for children and adolescents (12 to 17 years) is used. The Hemo-QoL-SF contains 35 questions covering 9 domains: Physical Health, View of Yourself, Family, Friends, Others, Sports, Dealing, and Treatment.
Changes of WPAI score | From baseline to 12 months, 24 months and 36 months
  WPAI:Work Productivity and Activity Impairment Scale。 Scores are expressed as percentages of impairment/ productivity loss, with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (10):
  - South Alabama Medical Science Foundation, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Phoenix, Arizona
  - University California Davis, Davis, California
  - Orthopaedic Hospital DBA Orthopaedic Institute for Children, Los Angeles, California
  - The Center for Comprehensive Care and Diagnosis of Inherited Blood Disorders, Orange, California
  - University of Colorado Hemophilia and Thrombosis Center, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Tulane University, New Orleans, Louisiana
  - Regents of University of Minnesota, Minneapolis, Minnesota
  - East Carolina University - Brody School of Medicine, Greenville, North Carolina
- Many locations, Multiple Locations, Belgium
- Many locations, Multiple Locations, Brazil
- Many locations, Multiple Locations, Canada
- Many locations, Multiple Locations, Colombia
- Many locations, Multiple Locations, Denmark
- Many locations, Multiple Locations, Germany
- Many locations, Multiple Locations, Greece
- Many locations, Multiple Locations, Italy
- Many locations, Multiple Locations, Japan
- Many locations, Multiple Locations, Kuwait
- Many locations, Multiple Locations, Netherlands
- Many locations, Multiple Locations, Norway
- Many locations, Multiple Locations, Saudi Arabia
- Many locations, Multiple Locations, Slovenia
- Many locations, Multiple Locations, Spain
- Many locations, Multiple Locations, Sweden
- Many locations, Multiple Locations, Switzerland
- Many locations, Multiple Locations, Taiwan
- Many locations, Multiple Locations, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Sanabria M, Alvarez Roman MT, Castaman G, Janbain M, Matsushita T, Meijer K, Oldenburg J, Friedl S, Reding MT. Design of the HEM-POWR study: a prospective, observational study of real-world treatment with damoctocog alfa pegol in patients with haemophilia A. BMJ Open. 2021 Sep 2;11(9):e044997. doi: 10.1136/bmjopen-2020-044997. PMID 34475142